CLINICAL TRIAL: NCT03098004
Title: Effects of Electronic Cigarettes on Nicotine Withdrawal Among Smokers
Brief Title: Effects of e-Cigarettes on Nicotine Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Adam Leventhal, Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HS-16-00630
Record Dates: First submitted 2017-03-22; First posted 2017-03-31 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Electronic Cigarettes
MeSH Terms: conditions — Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sweet-Flavored e-Cigarette (Experimental): Participants will self-administer a sweet-flavored e-cigarette containing 3 mg/mL of nicotine.
  Interventions: Other: e-Cigarette
- Tobacco-Flavored e-Cigarette (Active Comparator): Participants will self-administer a tobacco-flavored e-cigarette containing 3 mg/mL of nicotine.
  Interventions: Other: e-Cigarette

INTERVENTIONS:
Other: e-Cigarette — Participants will self-administer an experimenter-provided e-cigarette.

SUMMARY:
This behavioral pharmacology laboratory experiment will assess whether sweet (vs. non-sweet) flavored e-cigarette solutions reduce tobacco withdrawal symptoms and motivation to smoke among 40 smokers interested in trying e-cigarettes (for the first time) following 16-hours of nicotine abstinence. The study's experimental design will provide evidence of the causal effects of e-cigarette flavorings on a putatively critical factor for determining whether smokers continue e-cigarette use after initial trial-the ability of a product to suppress withdrawal and motivation to smoke during periods of tobacco deprivation.

DETAILED DESCRIPTION:
Nicotine withdrawal symptoms (e.g., increased negative affect, decreased positive affect, cigarette craving) are a core component of cigarette dependence that emerge upon the absence of nicotine administration, maintaining cigarette smoking and inhibiting cessation efforts. The use of electronic cigarettes (e-cigarettes) has increased dramatically in recent years, with studies demonstrating that e-cigarettes can reduce nicotine withdrawal symptoms during acute cigarette abstinence. E-cigarettes with flavorings that simulate the sweet taste of fruit, candy and other sugary foods and beverages are widely available, commonly used and are frequently cited as a reason for the persistent use of e-cigarettes. During nicotine withdrawal, sweet flavors have been shown to reduce nicotine withdrawal symptoms. Additionally, a recent USC TCORS (Tobacco Center of Regulatory Science) administrative supplement study conducted at the University of Southern California (USC) Health, Emotion, and Addiction Laboratory (USC-HEAL) found that sweet-flavored solutions enhanced the appeal of e-cigarettes, independent of nicotine. However, the impact of e-cigarette flavorings on nicotine withdrawal symptoms is currently unknown. This behavioral pharmacology laboratory experiment will assess whether sweet (vs. non-sweet) flavored e-cigarette solutions reduce tobacco withdrawal symptoms and motivation to smoke among 40 smokers interested in trying e-cigarettes (for the first time) following 16-hours of nicotine abstinence. At each visit, participants will complete a standardized e-cigarette administration procedure, as developed in our prior work, in which flavor will be manipulated in a double-blind, cross-over, counterbalanced design. Following the e-cigarette administration, participants will complete: 1) self-report measures of nicotine withdrawal symptoms; 2) physiological measurements and 3) a behavioral task that measures participants' ability to resist the desire to resume smoking under conditions in which it is advantageous to remain abstinent (i.e., monetary payment for each successive 5-min increment in which smoking is delayed). The study's experimental design will provide evidence of the causal effects of e-cigarette flavorings on a putatively critical factor for determining whether smokers continue e-cigarette use after initial trial-the ability of a product to suppress withdrawal and motivation to smoke during periods of tobacco deprivation.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years of age or older;
2. Daily cigarette smoking for at least the past two years;
3. Currently smoke > 10 cig/day;
4. Interest in trying e-cigarettes;
5. report primarily smoking non-mentholated cigarettes.

Exclusion Criteria:

1. Current use of medications that impact withdrawal or smoking (e.g., bupropion, varenicline, nicotine replacement, anti-depressants, anxiolytics);
2. Prior use of e-cigarettes (i.e., self-report > 10 puffs lifetime, use on more than two occasions, purchased own device);
3. breath carbon monoxide (CO) < 10 at intake;
4. pregnancy/breastfeeding; and
5. daily use of other tobacco products (e.g., hookah, cigars).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Positive Affect Negative Affect Schedule | 4 hours
  The 10-item Positive Affect Negative Affect Schedule (PANAS-SF) will be used to measure positive and negative affect.
The Minnesota Nicotine withdrawal Scale | 4 hours
  The Minnesota Nicotine withdrawal Scale (MNWS) measures 11 nicotine withdrawal symptoms on 6-point response scales.

SECONDARY OUTCOMES:
Wisconsin Smoking Withdrawal Scale | 4 hours
  Additional withdrawal symptoms (e.g., hunger, concentration problems) will be measured with the Wisconsin Smoking Withdrawal Scale (WSWS).
Questionnaire of Smoking Urges | 4 hours
  10-item Brief Questionnaire of Smoking Urges will assess desire, intention, urge and need to smoke cigarettes.

CONTACTS AND LOCATIONS:
Locations (1):
- USC Health, Emotion and Addiction Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No